CLINICAL TRIAL: NCT06805916
Title: Promoting Communicative Initiative in Minimally Verbal Autistic Children Through Interaction with the Humanoid Social Robot
Brief Title: Promoting Communication in Minimally Verbal Autistic Children with Social Robot
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Francesca Cucinotta, Principal Investigator, IRCCS Centro Neurolesi Bonino Pulejo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NAO01
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NAO-Assisted Intervention (Experimental Group EG) (Experimental): The treatment group consists of 50 children diagnosed with Autism Spectrum Disorder (ASD) who are minimally verbal (MV). Participants were randomly assigned and underwent a structured rehabilitative program integrated with the use of the NAO humanoid robot. The intervention was tailored to individual needs and aimed at improving communicative initiative, verbalization, and social engagement. Each child received therapy over a period of 12 weeks, totaling 12 sessions, once per week, with each session lasting 45 minutes.
  Interventions: Behavioral: NAO-Assisted Therapy
- Standard Therapy (Control Group) (Active Comparator): The control group consists of 50 children diagnosed with Autism Spectrum Disorder (ASD) who are minimally verbal (MV). Participants were randomly assigned and underwent standard therapeutic approaches, which included traditional speech therapy provided by trained therapists. The therapy followed established protocols and was adapted to meet the specific needs of minimally verbal children. Each child received therapy over a period of 12 weeks, totaling 12 sessions, once per week, with each session lasting 45 minutes.
  Interventions: Behavioral: Standard therapeutic

INTERVENTIONS:
Behavioral: NAO-Assisted Therapy — The intervention sessions included tasks designed to engage the child in verbal and social interactions, such as naming objects, responding to questions, and performing gestures. The NAO robot provided consistent and predictable feedback, while therapists supported and reinforced appropriate communicative behaviors.
  Arms: NAO-Assisted Intervention (Experimental Group EG)
Behavioral: Standard therapeutic — Standard therapeutic approaches included exercises aimed at improving verbal communication and social engagement, such as naming objects, sentence construction, and comprehension tasks. Therapists adapted the intervention to the child's individual communication goals.
  Arms: Standard Therapy (Control Group)

SUMMARY:
Minimally verbal (MV) children with Autism Spectrum Disorder (ASD) face significant challenges in communication and social interaction, which are fundamental to learning and development. Current therapeutic approaches, such as speech therapy and augmentative communication systems, often have variable efficacy due to engagement and responsiveness challenges. This pilot study investigates using of the humanoid robot NAO as part of a rehabilitative program designed for MV children with ASD. NAO, with its predictable and engaging interaction style, is hypothesized to enhance communicative initiative, expressive communication, and social interaction in this population. The study employs a randomized controlled trial design, assigning participants to either an NAO-assisted intervention group or a control group receiving standard therapy. Outcomes will be assessed using standardized measures of communication, social interaction, and observational data. This research aims to explore the potential of social robots as an innovative tool to addressing the unique needs of MV children with ASD, contributing to the development of effective, accessible therapeutic options that improve their quality of life and that of their families.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a complex neurodevelopmental condition characterized by deficits in social communication and restricted, repetitive patterns of behavior, interests, or activities. Among individuals with ASD, approximately 25-30% are minimally verbal (MV), demonstrating limited verbal or non-verbal communication skills, which poses significant challenges for social interaction and learning. Early diagnosis and tailored therapeutic interventions are crucial for improving long-term outcomes in this population. However, traditional therapies often face limitations, including variability in efficacy and difficulty maintaining engagement among MV children. In recent years, the integration of advanced technologies into therapeutic programs has gained traction as an innovative approach to address communication challenges in ASD. Social robots, such as the humanoid robot NAO, offer unique opportunities to engage children with ASD through consistent and predictable interactions. NAO is equipped with capabilities including speech recognition, gestures, and responses to touch and movement, making it an effective tool for promoting communication and social behaviors. Preliminary studies suggest that social robots can enhance engagement and improve social skills in children with ASD, yet their potential remains underexplored in minimally verbal children. This single-blind, randomized, controlled study aims to evaluate the feasibility and effectiveness of a rehabilitative treatment program integrating the NAO robot for minimally verbal children with ASD. NAO-assisted therapy sessions are designed to promote communicative initiative, expressive language, and social interaction through interactive tasks tailored to each child's needs.

The study's outcomes will be measured using standardized communication assessments, including the Test of Verbalization (TVL), and observational data to evaluate engagement, responsiveness, and frequency of communicative behaviors. By leveraging advanced robotic technology, this study aims to explore new avenues for therapeutic interventions, ultimately contributing to the development of evidence-based strategies that improve the quality of life for minimally verbal children with ASD and their families.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD)
* Minimal verbal communication
* Age between 4 and 12 years.

Exclusion Criteria:

* Presence of severe intellectual disability.
* Diagnosis of neurological disorders other than ASD.
* Significant medical conditions that could interfere with study participation.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Language Development Level Test (TVL) | T0(baseline)-T1(3months)
  The Test of Verbalization and Language Development (TVL) is a standardized tool designed to assess various aspects of language development, including verbal production, comprehension, sentence construction, phonological accuracy, and morphosyntactic abilities. The weighted score ranges from 0 to 10, with higher scores indicating better language development.
The Child Behavior Checklist (CBCL) | T0(baseline)-T1(3months)
  The Child Behavior Checklist (CBCL) is a caregiver-reported questionnaire used to identify emotional and behavioral problems in children. It measures multiple domains, including emotional reactivity, anxiety, attention problems, and social difficulties. The T-scores do not have a specific range, but values between 50 and 70 are considered within the normal range, while 70 to 100 indicates clinical significance. Higher scores indicate greater behavioral problems.
Quality of Life in Autism Questionnaire (QoLA) | T0(baseline)-T1(3months)
  The Quality of Life in Autism Questionnaire (QoLA) is a standardized measure assessing the quality of life of parents of autistic children, focusing on emotional well-being, stress, and satisfaction with support services. The questionnaire consists of two parts:
  * Part A: Scores range from 28 to 140, with higher scores indicating a better perceived quality of life.
  * Part B: Scores range from 20 to 100, with higher scores indicating fewer problems for parents related to their child's ASD-related behaviors.
Repetitive Behavior Scale (RBS) | T0(baseline)-T1(3months)
  The Repetitive Behavior Scale-Revised (RBS-R) is a caregiver-reported questionnaire assessing restricted and repetitive behaviors in autistic children, including stereotyped behaviors, self-injury, and compulsive behaviors. Each behavior is rated on a 4-point Likert scale. Higher scores indicate greater severity of repetitive behaviors.
Strengths and Difficulties Questionnaire (SDQ) | T0(baseline)-T1(3months)
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioral screening tool assessing emotional symptoms, conduct problems, hyperactivity, peer relationship problems, and prosocial behaviors in children aged 2-17 years.
  For all scales except the prosocial behavior scale, higher scores indicate greater levels of distress. In the prosocial behavior scale, higher scores indicate stronger positive social behaviors.
Conners' Parent Rating Scale (CPRS) | T0(baseline)-T1(3months)
  The Conners' Parent Rating Scale (CPRS) is a widely used research and clinical tool that gathers parental reports on childhood behavioral problems, particularly related to attention-deficit/hyperactivity disorder (ADHD) and associated behavioral concerns. T-scores above 70 indicate a higher likelihood of problematic behaviors and ADHD symptoms. Higher scores suggest greater severity of behavioral issues
Mand Requests During Sessions | During Sessions
  This observational measure tracks and records the number of spontaneous and prompted requests initiated by the child to express needs or desires during therapy sessions. Frequency count per session. Higher frequencies indicate greater communicative initiative

CONTACTS AND LOCATIONS:
Overall Officials: Margherita La Fauci, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo; Maria Tresoldi, Principal Investigator — University Hospital "G. Martino"; Marcella Di Cara, Principal Investigator — IRCCS Centro Neurolesi Bonino Pulejo
Locations (1):
- IRCCS Centro Neurolesi Bonino Pulejo, Messina, Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillingham KK, Makalous DL, Tays MA. G stress on A-10 pilots during JAWS II exercises. Aviat Space Environ Med. 1982 Apr;53(4):336-41. PMID 7082249
- [Background] Rose V, Trembath D, Keen D, Paynter J. The proportion of minimally verbal children with autism spectrum disorder in a community-based early intervention programme. J Intellect Disabil Res. 2016 May;60(5):464-77. doi: 10.1111/jir.12284. PMID 27120989
- [Background] Rybka J, Novosad P. Reaction of human organism to exercise. III. Biochemical response to physical loading. Acta Univ Carol Med (Praha). 1984;30(5-6):387-441. No abstract available. PMID 6516977
- [Background] Korneder J, Louie WG, Pawluk CM, Abbas I, Brys M, Rooney F. Robot-mediated interventions for teaching children with ASD: A new intraverbal skill. Assist Technol. 2022 Nov 2;34(6):707-716. doi: 10.1080/10400435.2021.1930284. Epub 2021 May 28. PMID 33983864
- [Background] Salimi Z, Jenabi E, Bashirian S. Are social robots ready yet to be used in care and therapy of autism spectrum disorder: A systematic review of randomized controlled trials. Neurosci Biobehav Rev. 2021 Oct;129:1-16. doi: 10.1016/j.neubiorev.2021.04.009. Epub 2021 Apr 20. PMID 33862066